CLINICAL TRIAL: NCT05965544
Title: The Effect of Application of Fascia Iliaca Compartment Block (FICB) Before or After Spinal Anesthesia on QoR-15 Score in Partial Hip Arthroplasty Surgery
Brief Title: The Effect of Fascia Iliaca Compartment Block (FICB) on QoR-15 Score in Partial Hip Arthroplasty Surgery
Acronym: QoR-15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Ergün Mendeş, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: e.mendes - 2; KAEK/2023.06.259 (Other: Basaksehir Cam and Sakura City Hospital)
Record Dates: First submitted 2023-07-13; First posted 2023-07-28 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Post Operative Pain; Anesthesia, Local; Fracture of Hip; QoR-15
Keywords: Fascia Iliaca Compartment Block; FICB; Partial Hip Arthroplasty Surgery; Quality of Recovery-15
MeSH Terms: conditions — Pain, Postoperative; Hip Fractures | interventions — Anesthesia, Spinal; Postoperative Period

STUDY DESIGN:
Intervention Model Description: The patients were equally randomized into two groups using a computer-generated random number table. In the preoperative period, according to whether FIBP was before or after spinal anesthesia, it was named as a separate group as Group PreS (Pre-Spinal) and Group PostS (Post-Spinal).
Who Masked: Care Provider, Outcomes Assessor
Masking Description: After each patient's eligibility has been assessed, numbered and sealed envelopes will be used to conceal assignment status. The same clinician (E.M.) will perform the patient's pre- and post-operative procedures. A researcher who does not know which method was applied to the patient in the perioperative and postoperative follow-ups will be included as double-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PreS (Active Comparator): The block will be applied in the preoperative period
  Interventions: Drug: Bupivacain (preoperative); Drug: Bupivacaine-fentanyl
- Group PostS (Active Comparator): The block will be applied in the postoperative period
  Interventions: Drug: Bupivacaine-fentanyl; Drug: Bupivacain (Postoperative)

INTERVENTIONS:
Drug: Bupivacain (preoperative) — After the patients are in the supine position and aseptic conditions are provided in the preoperative period, the fascia on the iliacus muscle will be determined with the help of an 8-12 MHz linear probe and a block will be applied with the in-plane technique. During the block, 0.2% bupivacaine concentration 0.5 mL/kg is routinely used in patients.
  Other Names: Preoperative Fascia Iliaca Compartment Block
  Arms: Group PreS
Drug: Bupivacaine-fentanyl — The patient will be placed in the lateral decubitus position with the fractured side up. After the spinal anesthesia method was provided with aseptic conditions, 10 mg 0.5% bupivacaine + 20 mcg Fentanyl injection will be applied using a 26 Gauge pencil point needle through the L3-L4 or L4-L5 intervertebral space
  Other Names: Spinal Anesthesia
Drug: Bupivacain (Postoperative) — After the patients are in the supine position and aseptic conditions are provided in the postoperative period, the fascia on the iliacus muscle will be determined with the help of an 8-12 MHz linear probe and a block will be applied with the in-plane technique. During the block, 0.2% bupivacaine concentration 0.5 mL/kg is routinely used in patients.
  Other Names: Postoperative Fascia Iliaca Compartment Block
  Arms: Group PostS

SUMMARY:
It reduces pain scores in patients with block and improves the quality of recovery in the postoperative period. In patients who will undergo spinal anesthesia, it will be questioned whether the application of the block before or after surgery makes a difference in the quality of recovery.

DETAILED DESCRIPTION:
American Society of Anesthesiologists (ASA) physical status I-III patients who are planned for partial hip arthroplasty will be studied in patients over 65 years of age. The patients will be equally randomized into two groups using a computer-generated random number table. In the preoperative period, according to whether FIBP was before or after spinal anesthesia, it will be named as a separate group as Group PreS (Pre-Spinal) and Group PostS (Post-Spinal). The patient will be placed in the lateral decubitus position with the fractured side up. After the spinal anesthesia method was provided with aseptic conditions, 10 mg 0.5% isobaric bupivacaine + 20 mcg Fentanyl injection will be applied using a 26 Gauge pencil point needle through the L3-L4 or L4-L5 intervertebral space. After the patients are in the supine position and aseptic conditions are provided, the fascia on the Iliacus muscle will be determined with the help of an 8-12 MHz linear probe, and the block will be applied with the in-plane technique. During the block, patients will routinely administer 0.2% bupivacaine concentration of 0.5 mL/kg. Demographic data, operation time, perioperative analgesic and sedation need, postoperative pain scores, additional analgesic need, hospitalization and 24th-hour recovery scores will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Partial Hip Arthroplasty
* American Society of Anesthesiologists (ASA) physical status I-III,
* Patients aged ≥ 65 years

Exclusion criteria:

* Contraindication for central or peripheral blocks,
* Cognitive Dysfunction,
* History of chronic opioid use,
* Previous hip surgery,
* Serious organ dysfunction,
* Allergy to any drug used in the study,
* Body mass index (BMI) ≥30,
* Infection in the area to be treated,
* Refusal to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline QoR-15 at 24 hours postoperatively | Postoperative 24th-hours
  The patient-reported Turkish QoR-15 score includes 15 questions that evaluate the patient's postoperative recovery. The QoR-15 score is grouped under two groups, A and B. A high QoR-15 score, a score between 0 (poor) and 10 (excellent) for each item, and a total score of 150 indicate better quality of recovery.

SECONDARY OUTCOMES:
Change from baseline Nursing Delirium Screening Scale (N-DSS) at 24 hours postoperatively | Postoperative 24th-hours
  Postoperative delirium will be determined with the Nursing Delirium Screening Scale (N-DSS), an easily applicable five-item screening tool that evaluates disorientation, inappropriate behavior, inappropriate communication, hallucination, and psychomotor retardation. Each item scores between 0 and 2 and the total score varies between 0 and 10.
Postoperative nausea and vomiting | Postoperative 24th hour
  The frequency of nausea and vomiting in the postoperative period was calculated according to the Numeric Rank Score (NRS), which ranged from 0 to 3. Nausea-vomiting status of the patients: 0 points if there is no nausea and vomiting; 1 point if there is nausea, no vomiting; It is scored as 2 points if there is vomiting once and 3 points if there are two or more vomiting attacks.
Analgesic consumption | Postoperative 24th hour
  The value in mg of the amount of analgesic consumed in the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Ergun Mendes, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Ergun Mendes, Küçükçekmece, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Selvi O, Azizoglu M, Temel G, Tulgar S, Chitneni A, Cinar EN, Ozer Z, Gurkan Y. Translation and Validation of the Turkish Version of the Quality of Postoperative Recovery Score QoR-15: A Multi-Centred Cohort Study. Turk J Anaesthesiol Reanim. 2022 Dec;50(6):443-448. doi: 10.5152/TJAR.2022.21417. PMID 36511494
- [Derived] Mendes E, Adiyeke O, Sarban O, Civan M, Ozcan FG. Timing of suprainguinal fascia iliaca block in hip hemiarthroplasty: impact on QoR-15 scores- a prospective randomized study. BMC Anesthesiol. 2025 Apr 12;25(1):179. doi: 10.1186/s12871-025-03060-8. PMID 40221676